CLINICAL TRIAL: NCT02992119
Title: Safety and Immunogenicity Evaluation of the Malaria Vaccine, RTS,S/AS01, in Healthy Thai Adults
Brief Title: Malaria Vaccine Safety and Immunogenicity Study in Healthy Adults
Acronym: RTSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAKMAL1605
Record Dates: First submitted 2016-11-15; First posted 2016-12-14 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2019-07

CONDITIONS: Malaria Vaccine
Keywords: safety; immunogenicity
MeSH Terms: interventions — RTS malaria vaccine

STUDY DESIGN:
Intervention Model Description: Randomized 7 groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1 (Experimental): RTS,S/AS01B Fractional dose
  Interventions: Biological: RTS,S/AS01B Fractional dose
- Group 2 (Experimental): Double RTS,S/AS01E Fractional dose
  Interventions: Biological: Double RTS,S/AS01E Fractional dose
- Group 3 (Experimental): RTS,S/AS01E Standard dose
  Interventions: Biological: RTS,S/AS01E Standard dose
- Group 4 (Experimental): RTS,S/AS01E + DHA-PIP+PQ Standard dose
  Interventions: Biological: RTS,S/AS01E + DHA-PIP+PQ Standard dose
- Group 5 (Experimental): RTS,S/AS01E Fractional dose
  Interventions: Biological: RTS,S/AS01E Fractional dose
- Group 6 (Experimental): RTS,S/AS01E + DHA-PIP+PQ Fractional dose
  Interventions: Biological: RTS,S/AS01E + DHA-PIP+PQ Fractional dose
- Group 7 (Experimental): RTS,S/AS01E + DHA-PIP+PQ Fractional two-dose
  Interventions: Biological: RTS,S/AS01E + DHA-PIP+PQ Fractional two-dose

INTERVENTIONS:
Biological: RTS,S/AS01B Fractional dose — RTS,S/AS01B standard dose at Month 0 and Month 1 + RTS,S/AS01B fractional dose (1/5th dose) at Month 2.
  Arms: Group 1
Biological: Double RTS,S/AS01E Fractional dose — A double dose of RTS,S/AS01E standard dose at Month 0 and Month 1 + a double dose of RTS,S/AS01E fractional dose (1/5th dose) at Month 2.
  Arms: Group 2
Biological: RTS,S/AS01E Standard dose — RTS,S/AS01E standard dose at Month 0, Month 1 and Month 2.
  Arms: Group 3
Biological: RTS,S/AS01E + DHA-PIP+PQ Standard dose — RTS,S/AS01E standard dose + DHA-PIP+PQ at Month 0, Month 1 and Month 2
  Arms: Group 4
Biological: RTS,S/AS01E Fractional dose — RTS,S/AS01E standard dose at Month 0 and Month 1 + RTS,S/AS01E fractional dose (1/5th dose) at Month 2.
  Arms: Group 5
Biological: RTS,S/AS01E + DHA-PIP+PQ Fractional dose — RTS,S/AS01E standard dose + DHA-PIP+PQ at Month 0 and Month 1 + RTS,S/AS01E fractional dose (1/5th dose) + DHA-PIP+PQ at Month 2.
  Arms: Group 6
Biological: RTS,S/AS01E + DHA-PIP+PQ Fractional two-dose — RTS,S/AS01E standard dose + DHA-PIP+PQ at Month 0 + RTS,S/AS01E fractional dose (1/5th dose) + DHA-PIP+PQ at Month 2
  Arms: Group 7

SUMMARY:
Targeted malaria elimination (TME), which comprises appropriate case management by village health workers, vector control and mass drug administration, is currently being implemented through pilot projects in selected villages in the Greater Mekong Subregion (GMS) and the scale-up of the intervention to the regional level are underway. Based on mathematical modelling, extending the post-TME parasitaemia-free period in the majority of villagers for as short as 200 days will substantially increase the chances of achieving the interruption of malaria transmission. Immunogenicity of RTS,S is greater in older children, and the short term malaria protective effect is stronger than the overall effect assessed over 1-2 years. Addition of mass RTS,S/AS01E vaccination to the TME arsenal could provide this much needed additional protection.

Currently there are no safety and immunogenicity data for the use of RTS,S/AS01 in Asian populations. This trial will generate the required data for the use of this vaccine in Asian populations. For integration with the current TME activities, which provide mass drug administrations at months M0, M1, and M2, it would be most efficient and practical to provide the vaccine at the same intervals. To address a two round intervention (M0, M2) where a three round intervention is not feasible, one study arm will look at the immune response generated by only two doses of vaccine and antimalarial medications. Recent evidence suggests that a vaccination schedule which includes a fractional dose of RTS,S/AS01 (1/5th of the standard dose) could be similarly or more protective than a schedule with three standard full doses, while requiring less vaccine and resources. The trial therefore includes study arms which will assess the safety and immunogenicity of fractional dose schedules.

Each participant will be randomized into one of the following study arms in a ratio of 20:20:30:30:30:30:30, as follows:

* RTS,S/AS01B Fractional dose group (Group 1)
* Double RTS,S /AS01E Fractional dose group (Group 2)
* RTS,S/AS01E Standard dose group (Group 3)
* RTS,S/AS01E + DHA-PIP+PQ Standard dose group (Group 4)
* RTS,S/AS01E Fractional dose group (Group 5)
* RTS,S/AS01E + DHA-PIP+PQ Fractional dose group (Group 6)
* RTS,S/AS01E + DHA-PIP+PQ Fractional two-dose group (Group 7)

DETAILED DESCRIPTION:
This is a randomized, open-label, single centre, Phase 2 trial of RTS,S/AS01 in healthy Thai adults.

Screening and eligibility assessment (Screening visit)

All potential volunteers will have a screening visit, which may take place up to 30 days prior to enrolment. Once informed consent is given, a screening number will be assigned in sequential order. Screening numbers will be issued consecutively (e.g. A-01, A-02, A-03…).

Enrolment, baseline assessment, regimen allocation, and first vaccination (Month 0 / Day 0 visit; Baseline visit) All inclusion and exclusion criteria will be checked before enrolment in the study. Physical examination will be performed. Any new medical issues or symptoms that have arisen will be assessed. Blood will be collected for baseline parasite microscopy, haemoglobin and biochemistry. Participants with parasitaemia or anaemia will be treated according to national guidelines. Blood will be collected and stored for measurement of antibodies against P. falciparum circumsporozoite (anti-CS antibody) until shipment to the reference laboratory. Urine will be collected from women of child-bearing age for immediate pregnancy test.

If all inclusion criteria are fulfilled and none of the exclusion criteria apply, the patient will be enrolled into the study and a CRF specific to each participant completed. Regimen allocation and administration of the vaccine(s) will be on Day 0. The randomization lists will be prepared by MORU.

Randomization numbers will be generated in blocks, for the 7 intervention arms in a ratio of 20:20:30:30:30:30:30, as follows:

Each participant will be randomized into one of the following study arms Group 1: RTS,S/AS01B Fractional dose group Month 0 and Month 1 will receive RTS,S/AS01B full dose Month 2 will receive RTS,S/AS01B fractional dose (1/5th dose)

Group 2: RTS,S/AS01E Fractional dose group Month 0 and Month 1will receive a double dose of RTS,S/AS01E full dose Month 2 will receive a double dose of RTS,S/AS01E fractional dose (1/5th dose)

Group 3: RTS,S/AS01E Full dose group Month 0, Month 1 and Month 2 will receive RTS,S/AS01E full dose

Group 4: RTS,S/AS01E + DHA-PIP+PQ Full dose group Month 0, Month 1 and Month 2 will receive RTS,S/AS01E full dose + DHA-PIP+PQ

Group 5: RTS,S/AS01E Fractional dose group Month 0 and Month 1 will receive RTS,S/AS01E full dose Month 2 will receive RTS,S/AS01E fractional dose (1/5th dose)

Group 6: RTS,S/AS01E + DHA-PIP+PQ Fractional dose group Month 0 and Month 1 will receive RTS,S/AS01E full dose + DHA-PIP+PQ Month 2 will receive RTS,S/AS01E fractional dose (1/5th dose) + DHA-PIP+PQ

Group 7: RTS,S/AS01E + DHA-PIP+PQ Fractional two-dose group Month 0 will receive RTS,S/AS01E full dose + DHA-PIP+PQ Month 2 will receive RTS,S/AS01E fractional dose (1/5th dose) + DHA-PIP+PQ

RTS,S/AS01B = Standard dose RTS,S/AS01B: 50µg RTS,S + standard dose AS01B RTS,S/AS01E = Standard dose RTS,S/AS01E: 25µg RTS,S + standard dose AS01E DHA-PIP = Dihydroartemisinin/piperaquine PQ = Primaquine

Study participants will be assigned the next available randomization number on the list, and thus will be randomly allocated to Group 1, 2, 3, 4, 5, 6 or 7.

Subsequent vaccination visits (Month 1 / Day 0 and Month 2 / Day 0 visits) Subsequent vaccination visits will be done according to the schedule of procedures. Physical examination will be performed. Any new medical issues or symptoms that have arisen will be assessed. Blood will be collected for parasite microscopy, haemoglobin and biochemistry. Participants with parasitaemia or anaemia will be treated according to national guidelines. Blood will be collected and stored for measurement of antibodies against P. falciparum circumsporozoite (anti-CS antibody) until shipment to the reference laboratory. Urine will be collected from women of child-bearing age for immediate pregnancy test.

Before vaccination, the on-going eligibility of the volunteer will be reviewed. All participants will attend the clinic for vaccination visits, will be observed closely for at least 30 minutes following the administration of each study vaccine, and will receive a paper diary card for recording solicited AEs, as described above. Information will be recorded in the CRF for subsequent vaccination visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a healthy male or non-pregnant female, aged 18 to 55 years (inclusive), of Thai origin.
* Participant is willing and able to give informed consent to participate in the trial
* Able, in the investigators opinion, and willing to comply with the study requirements and follow-up.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Presence of any condition which in the judgment of the investigator would place the participant at undue risk or interfere with the results of the study (e.g. serious underlying cardiac, renal, hepatic or neurological disease; severe malnutrition; congenital defects or febrile condition).
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Screening ECG demonstrates a QTc interval ≥ 450 ms
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Anaemia (Hb < 10 g/dL)
* Positive malaria parasitaemia at screening or baseline (Month 0, Day 0).
* Use of any investigational or non-registered product or investigational use of a registered product (drug or vaccine), other than the study vaccines, during the period from the date of screening to the first vaccination, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular (IM) injection unsafe.
* Any medical condition that in the judgment of the investigator would make the administration of the antimalarial treatment unsafe, such as prior allergic reactions to one or more component of the drug regimen: artemisinins, piperaquine or primaquine.
* Contraindications to the use of artemisinins, piperaquine or primaquine or use of medications known to have a potentially clinically significant interaction with these medications.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone > 20 mg/day (for adult subjects), or equivalent. Inhaled and topical steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting seven days before the first dose.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* History of splenectomy.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection or based on medical history and physical examination.
* History of anaphylaxis post-vaccination.
* Serious chronic illness.
* Any abnormal baseline laboratory screening tests: ALT, AST, creatinine, haemoglobin, platelet count, total WBC, out of normal range as defined in the protocol.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Personal history of autoimmune disease.
* Administration of immunoglobulins and/or any blood products during the period starting three months before the first dose of study vaccine or planned administration during the study period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2017-06-04 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz von Seidlein, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Hospital of Tropical Diseases, Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 RTS,S/AS01B Fractional Dose: RTS,S/AS01B Fractional dose
  RTS,S/AS01B Fractional dose: RTS,S/AS01B standard dose at Month 0 and Month 1 + RTS,S/AS01B fractional dose (1/5th dose) at Month 2.
- Group 2 Double RTS,S/AS01E Fractional Dose: Double RTS,S/AS01E Fractional dose
  Double RTS,S/AS01E Fractional dose: A double dose of RTS,S/AS01E standard dose at Month 0 and Month 1 + a double dose of RTS,S/AS01E fractional dose (1/5th dose) at Month 2.
- Group 3 RTS,S/AS01E Standard Dose: RTS,S/AS01E Standard dose
  RTS,S/AS01E Standard dose: RTS,S/AS01E standard dose at Month 0, Month 1 and Month 2.
- Group 4 RTS,S/AS01E + DHA-PIP+PQ Standard Dose: RTS,S/AS01E + DHA-PIP+PQ Standard dose
  RTS,S/AS01E + DHA-PIP+PQ Standard dose: RTS,S/AS01E standard dose + DHA-PIP+PQ at Month 0, Month 1 and Month 2
- Group 5 RTS,S/AS01E Fractional Dose: RTS,S/AS01E Fractional dose
  RTS,S/AS01E Fractional dose: RTS,S/AS01E standard dose at Month 0 and Month 1 + RTS,S/AS01E fractional dose (1/5th dose) at Month 2.
- Group 6 RTS,S/AS01E + DHA-PIP+PQ Fractional Dose: RTS,S/AS01E + DHA-PIP+PQ Fractional dose
  RTS,S/AS01E + DHA-PIP+PQ Fractional dose: RTS,S/AS01E standard dose + DHA-PIP+PQ at Month 0 and Month 1 + RTS,S/AS01E fractional dose (1/5th dose) + DHA-PIP+PQ at Month 2.
- Group 7 RTS,S/AS01E + DHA-PIP+PQ Fractional Two-dose: RTS,S/AS01E + DHA-PIP+PQ Fractional two-dose
  RTS,S/AS01E + DHA-PIP+PQ Fractional two-dose: RTS,S/AS01E standard dose + DHA-PIP+PQ at Month 0 + RTS,S/AS01E fractional dose (1/5th dose) + DHA-PIP+PQ at Month 2
Period: Overall Study
Arm/Group | Group 1 RTS,S/AS01B Fractional Dose | Group 2 Double RTS,S/AS01E Fractional Dose | Group 3 RTS,S/AS01E Standard Dose | Group 4 RTS,S/AS01E + DHA-PIP+PQ Standard Dose | Group 5 RTS,S/AS01E Fractional Dose | Group 6 RTS,S/AS01E + DHA-PIP+PQ Fractional Dose | Group 7 RTS,S/AS01E + DHA-PIP+PQ Fractional Two-dose
Started | 21 | 21 | 30 | 30 | 30 | 30 | 31
Completed | 19 | 20 | 29 | 30 | 30 | 30 | 28
Not Completed | 2 | 1 | 1 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7 | Total
Number analyzed (Participants) | 21 | 21 | 30 | 30 | 30 | 30 | 31 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 30 | 30 | 30 | 30 | 31 | 193
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 16 | 17 | 17 | 16 | 17 | 106
  Male | 9 | 10 | 14 | 13 | 13 | 14 | 14 | 87
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
fever [Count of Participants; unit: Participants] — Fever is defined as temperature >= 37.5°C / 99.5°F for oral, axillary or tympanic route, or >= 38.0°C / 100.4°F for rectal route. The preferred route for recording temperature in this study will be oral.
  For subjects self temperature recording at home, they were instructed to record temperature in the evening time. Population: Analysed all participants at the baseline visit
  Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience a Serious Adverse Events (SAEs) 29 Days After the Last Vaccination
Description: Occurrence of serious adverse events (SAEs) from the date of the first vaccination to 29 days after the last vaccination, according to the MedRA classification.
Time Frame: 29 days after last vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 19 | 20 | 29 | 30 | 30 | 30 | 28
Participants | 1 | 0 | 0 | 1 | 1 | 0 | 0

2. Primary Outcome: Number of Participants Who Experience a Serious Adverse Events (SAEs) During a 6 Month Follow up Period From the Receipt of First Vaccination
Description: Occurrence of SAEs during the whole study period, i.e. during a 6 month follow up period from the receipt of first vaccination, according to the MedRA classification.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 21 | 21 | 30 | 30 | 30 | 30 | 31
Participants | 1 | 0 | 0 | 1 | 1 | 0 | 0

3. Primary Outcome: Number of Participants Who Seroconverted One Month After First Dose.
Description: The percentage of subjects seroconverting after each immunization based on a value greater than the mean titer at baseline (before immunization # 1) plus 2 standard deviations for all subjects included in the analysis (ITT).
Time Frame: 1 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 20 | 20 | 30 | 30 | 30 | 30 | 30
Participants | 20 | 20 | 29 | 30 | 28 | 29 | 30

4. Primary Outcome: Number of Participants Who Seroconverted One Month After the Second Dose.
Description: as for outcome 3
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6
Number analyzed (Participants) | 20 | 20 | 30 | 30 | 30 | 30
Participants | 19 | 20 | 30 | 30 | 30 | 30

5. Primary Outcome: Number of Participants Who Seroconverted One Month After the Third Dose.
Description: as for outcome 3
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 20 | 20 | 30 | 30 | 30 | 30 | 30
Participants | 20 | 20 | 30 | 30 | 30 | 30 | 30

6. Primary Outcome: Number of Participants Who Seroconverted at Month Six After First Dose.
Description: as for outcome 3
Time Frame: 6 months
Population: Analysed subjects who returned for the month 6 follow-up.
  There are 4 subjects lost follow-up as follows:
  1 subject from group 1
  1. subject from group 3
  2. subjects from group 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
Number analyzed (Participants) | 19 | 20 | 29 | 30 | 30 | 30 | 28
Participants | 19 | 20 | 29 | 30 | 30 | 30 | 27

7. Primary Outcome: Number of Participants Who Received RTS,S/AS01E + DHA-PIP+PQ Fractional Two-dose (Group 7) That Seroconverted at Month Two After First Dose.
Description: The percentage of subjects seroconverting after each immunization based on a value greater than the mean titer at baseline (before immunization # 1) plus 2 standard deviations for all subjects included in the analysis (ITT).(For group 7)
Time Frame: 2 months
Population: There were 30 subjects at group 7 received 1st vaccination and came back for follow-up at month 2 visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 7
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: 6 months
Description: clinicaltrials.gov definitions
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Group 6 | Group 7
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/30 | 0/30 | 0/30 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21 | 0/30 | 1/30 | 1/30 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 21/21 | 21/21 | 30/30 | 29/30 | 30/30 | 29/30 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=21) | Group 2 (N=21) | Group 3 (N=30) | Group 4 (N=30) | Group 5 (N=30) | Group 6 (N=30) | Group 7 (N=31)
acute pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 0 | 1 (1) | 0 (0) | 0 | 0
Depression (Psychiatric disorders) | 1 (1) | 0 | 0 | 0 (0) | 0 (0) | 0 | 0
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 0 | 0 (0) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=21) | Group 2 (N=21) | Group 3 (N=30) | Group 4 (N=30) | Group 5 (N=30) | Group 6 (N=30) | Group 7 (N=31)
Injection site pain (Injury, poisoning and procedural complications) | 20 (46) | 20 (42) | 30 (79) | 25 (60) | 29 (65) | 27 (57) | 28 (48)
Fatigue (General disorders) | 18 (41) | 16 (23) | 24 (53) | 21 (44) | 19 (34) | 25 (56) | 19 (31)
Headache (Nervous system disorders) | 14 (27) | 13 (17) | 19 (42) | 14 (23) | 14 (20) | 17 (29) | 11 (17)
Pyrexia (General disorders) | 13 (18) | 13 (19) | 16 (22) | 14 (21) | 12 (18) | 16 (22) | 8 (9)
Malaise (General disorders) | 9 (15) | 5 (7) | 8 (12) | 11 (15) | 5 (5) | 14 (15) | 8 (9)
Injection site reaction (pain) (Injury, poisoning and procedural complications) | 8 (14) | 6 (10) | 9 (18) | 6 (10) | 8 (16) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (4) | 3 (6) | 12 (22) | 3 (5) | 6 (8) | 4 (7)
Injection site reaction (redness) (Injury, poisoning and procedural complications) | 2 (3) | 10 (14) | 7 (14) | 3 (7) | 6 (10) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3) | 2 (4) | 4 (6) | 4 (5) | 8 (15) | 3 (4)
Haemoglobin low (General disorders) | 2 (2) | 1 (1) | 7 (7) | 6 (6) | 3 (3) | 4 (4) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (9) | 2 (3) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 3 (3) | 4 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 8 (8) | 2 (2) | 5 (5) | 3 (4)
Loose stools (Investigations) | 0 (0) | 0 (0) | 4 (4) | 6 (6) | 0 (0) | 1 (1) | 7 (7)
chills (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 4 (4) | 5 (5) | 1 (1) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT02992119/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT02992119/SAP_001.pdf